CLINICAL TRIAL: NCT04083378
Title: Clinical Impact of a Volumetric Image Method for Confirming Tumor Coverage With Ablation on Patients With Malignant Liver Lesions (COVER-ALL)
Brief Title: Software-Aided Imaging (Morfeus) for Confirming Tumor Coverage With Ablation in Patients With Liver Tumors, the COVER-ALL Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0213; NCI-2019-05762 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0213 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Malignant Liver Neoplasm
MeSH Terms: interventions — Catheter Ablation; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care ablation) (Active Comparator): Patients undergo standard of care ablation.
  Interventions: Procedure: Ablation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (standard of care ablation, software-aided imaging) (Experimental): Patients undergo standard of care ablation with software-aided imaging (Morfeus).
  Interventions: Procedure: Ablation Therapy; Procedure: Image-Guided Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Ablation Therapy — Undergo standard of care ablation
  Other Names: ABLATION; Catheter Ablation; Local Ablation Therapy; Local Ablative Therapy
Procedure: Image-Guided Therapy — Undergo software-aided imaging (Morfeus)
  Other Names: Image Guided Therapy; Imaging Guided Therapy
  Arms: Arm II (standard of care ablation, software-aided imaging)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well software-aided imaging works in confirming tumor coverage with ablation (the removal or destruction of a body part or tissue or its function) on patients with liver tumors. The current standard for targeting tumor cells and evaluating the outcome of a liver ablation procedure is a visual inspection of the pre- and post-procedure computed tomography (CT) scans. Software-aided imaging systems, such as Morfeus, may help to improve the accuracy and effectiveness of liver ablation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate if the intra-procedure feedback of a biomechanical deformable registration volumetric image method during percutaneous ablation will increase the minimal ablation margins on a three-dimensional computed tomography-generated analysis.

SECONDARY OBJECTIVES:

I. To assess whether applying the proposed method during percutaneous ablation improves local tumor progression-free survival (LTPFS) rates.

II. Evaluate impact of software use on procedure workflow.

III. Impact of software use on complication rates, quality of life, liver function.

IV. Evaluate oncological outcomes (intra-hepatic and overall progression-free survivals, and overall survival).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo standard of care ablation.

ARM II: Patients undergo standard of care ablation with software-aided imaging (Morfeus).

After completion of study, patients are followed up at 1, 3, and 6 months, and then at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with ≤ 3 liver tumors (biopsy-proven or documented by imaging) measuring 1 to 5 cm planned to undergo percutaneous thermal ablation with either microwave or radiofrequency ablation. Patients with more than 3 tumors might also be eligible in case other tumors can be treated with another curative-intended loco-regional therapy (i.e. surgical resection, radiation therapy).
2. Ability to completely cover the target tumor with at least a 5 mm ablation margin.
3. Written informed consent to voluntarily participate in the study and follow-up CT scan schedule
4. Age > 18 years-old
5. Performance status 0-2 (Eastern Cooperative Oncology Group Classification [ECOG])
6. Target tumor should be visualized on contrast-enhanced CT
7. Adequate glomerular filtration rate

Exclusion Criteria

1. Active bacterial infection or fungal infection on the day of the ablation that, in the opinion of the investigator, would interfere with safe delivery of the study procedure or with the interpretation of study results.
2. Platelet < 50,000/mm3.
3. INR > 1.5
4. Patients with uncorrectable coagulopathy.
5. Currently breastfeeding or pregnant (latter confirmed by serum pregnancy test).
6. Physical or psychological condition which would impair study participation.
7. ASA (American Society of Anesthesiologists) score of > 4.
8. Any other loco-regional therapies at the target lesion(s) within 30 days of the ablation procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2026-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: BRUNO C ODISIO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Odisio BC, Albuquerque J, Lin YM, Anderson BM, O'Connor CS, Rigaud B, Briones-Dimayuga M, Jones AK, Fellman BM, Huang SY, Kuban J, Metwalli ZA, Sheth R, Habibollahi P, Patel M, Shah KY, Cox VL, Kang HC, Morris VK, Kopetz S, Javle MM, Kaseb A, Tzeng CW, Cao HT, Newhook T, Chun YS, Vauthey JN, Gupta S, Paolucci I, Brock KK. Software-based versus visual assessment of the minimal ablative margin in patients with liver tumours undergoing percutaneous thermal ablation (COVER-ALL): a randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2025 May;10(5):442-451. doi: 10.1016/S2468-1253(25)00024-X. Epub 2025 Mar 13. PMID 40090348
- [Derived] Lin YM, Paolucci I, Anderson BM, O'Connor CS, Rigaud B, Briones-Dimayuga M, Jones KA, Brock KK, Fellman BM, Odisio BC. Study Protocol COVER-ALL: Clinical Impact of a Volumetric Image Method for Confirming Tumour Coverage with Ablation on Patients with Malignant Liver Lesions. Cardiovasc Intervent Radiol. 2022 Dec;45(12):1860-1867. doi: 10.1007/s00270-022-03255-3. Epub 2022 Sep 4. PMID 36058995
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: MD Anderson Cancer Center
Pre-assignment Details: Randomized and non-randomized experimental groups were combined as both received the same ablation confirmation (AC) software. Per DSMB recommendation, an interim stopping rule for control enrollment, which was triggered, halting further accrual. Thus, analyses comparing experimental versus control are presented in this simplified structure to ensure consistency in evaluating the novel AC software for liver tumor ablation.
Groups:
- Experimental: Clinical impact of Morfeus software usage on patients undergoing percutaneous ablation of hepatic mets
- Control: Morfeus software was not used during percutaneous ablation of hepatic mets
Period: Overall Study
Arm/Group | Experimental | Control
Started | 74 | 26
Completed | 52 | 22
Not Completed | 22 | 4
Not completed — Death | 18 | 4
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Population: Randomized and non-randomized experimental groups were combined as both received the same ablation confirmation (AC) software. Per DSMB recommendation, an interim stopping rule for control enrollment, which was triggered, halting further accrual. Thus, analyses comparing experimental versus control are presented in this simplified structure to ensure consistency in evaluating the novel AC software for liver tumor ablation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 74 | 26 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 18 | 70
  >=65 years | 22 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 8 | 39
  Male | 43 | 18 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 69 | 20 | 89
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 1 | 5
  White | 57 | 18 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 74 | 26 | 100

OUTCOME MEASURES:

1. Primary Outcome: Minimal Ablative Margin Assessment on Post-ablation Intraprocedural CT.
Description: For control group, MAM was assessed by rigid co-registration with side-by-side juxtaposition to verify applicator placement and by visual landmark-based CT measurements on CT workstation (Siemens Healthineers; Forchheim, Germany). For experimental group, CT images were processed with a software-based method on a radiation treatment planning system (Raystation, RaySearch Laboratories; Stockholm, Sweden) with biomechanical deformable imaging registration coupled with AI-based autosegmentation. For experimental group, interventional radiologist (IR) was informed of ablation applicator position relative to tumor on non-contrast CT before thermal ablation energy delivery and of MAM results (including spatial location of suboptimal margins) generated by software-based assessment, with this information not disclosed to IR in control group. Software-based assessment was used to compare MAMs results between both study groups with a two-sample t-test.
Time Frame: Visit 2 (baseline/ablation day)
Population: The primary endpoint included all enrolled patients
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Experimental: Clinical impact of Morfeus software usage on patients undergoing percutaneous ablation of liver tumors
- Control: Morfeus software was not used during percutaneous ablation of liver tumors
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 26
mm | 6.8 (2.9) | 2.2 (2.8)

2. Secondary Outcome: Cumulative Incidence of 2-year Local Tumor Progression
Description: A competing risk analysis was conducted to estimate the 2-year cumulative incidence of local tumor progression. Progression followed ablation reporting standards and RECIST v1.1 (mRECIST for HCC).
Time Frame: Time to local tumor progression (LTP) was measured from ablation to earliest LTP or death (competing event). Follow-up imaging continued up to 24 months.
Population: The 2-year secondary endpoints were evaluated for the randomized group
Measure: Number; unit: percentage of participants
Groups:
- Experimental: Clinical impact of Morfeus software usage on patients undergoing percutaneous thermal ablation of liver tumors
- Control: Morfeus software was not used during percutaneous thermal ablation of liver tumors
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 26
percentage of participants | 6 | 17.9

3. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method was used to estimate overall survival
Time Frame: Overall survival was measured from the date of ablation to the date of death from any cause. Patients still alive were censored at the date of last clinic visit, with follow-up up to 24 months after ablation.
Population: The 2-year secondary endpoints were evaluated for the randomized group
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 26
percentage of participants | 73.9 [64.2 to 85.0] | 83.6 [70.1 to 99.7]

4. Secondary Outcome: Intrahepatic Progression-free Survival (for the Randomized Group)
Description: Competing risk analysis was conducted to estimate the 2-year intrahepatic (progression outside of ablation zone), considering the progression of the ablated tumor and treating death as a competing event.
Time Frame: Up to 2 years
Population: The 2-year secondary endpoints are provided in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 26
percentage of participants | 34.5 [24.8 to 47.8] | 41.4 [25.4 to 67.3]

5. Secondary Outcome: Extrahepatic Progression-free Survival
Description: Competing risk analysis was conducted to estimate the 2-year extrahepatic cumulative incidence of progression, considering the progression of the ablated tumor and treating death as a competing event.
Time Frame: Up to 2 years
Population: The 2-year secondary endpoints are provided in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 26
percentage of participants | 34.5 [24.8 to 47.8] | 41.4 [25.4 to 67.3]

ADVERSE EVENTS:
Time Frame: Enrollment to 2-year follow-up, lost of follow-up, or death, whichever occurred first. AEs were classified as related (within 30 days) and unrelated to the thermal ablation procedure.
Description: Post-ablation syndrome (PAS) is a common, self-limited adverse event (AE) after thermal ablation, marked by transient fever, fatigue, leukocytosis, and flu-like symptoms within 24-72 h, resolving in 7-10 days. AEs related to PAS were recorded as per CTCAE v5.0 within 30 days of ablation and not specifically labeled as PAS.
Groups:
- Control: Morfeus software was not used during the percutaneous ablation of liver tumors
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 26/74 | 6/26
Serious Adverse Events (participants affected / at risk) | 39/74 | 12/26
Other Adverse Events (participants affected / at risk) | 18/74 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=74) | Control (N=26)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Allergic reaction (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Breast infection (Infections and infestations) | 1 (1) | 0 (0)
Bleeding (Vascular disorders) | 2 (2) | 0 (0)
Death (General disorders) | 26 (26) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dehydration (General disorders) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Encephalopathy (liver) (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (hip) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infection (suspected cholangitis) (Infections and infestations) | 1 (1) | 0 (0)
Ischemia (vascular disorder) (Vascular disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding (vaginal) (Vascular disorders) | 1 (1) | 0 (0)
Infection (Urinary Tract) (Infections and infestations) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Creatinine increased (Investigations) | 1 | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=74) | Control (N=26)
Abdominal pain (Gastrointestinal disorders) | 5 (12) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (COVID-19) (Infections and infestations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Rectal pain (General disorders) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT04083378/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT04083378/ICF_000.pdf